CLINICAL TRIAL: NCT01082250
Title: AN OPEN-LABEL, RANDOMIZED, THREE-PERIOD, TWO-SEQUENCE CROSSOVER, REPEATED-DOSE, REPLICATE DESIGN STUDY TO DETERMINE THE BIOEQUIVALENCE OF TWO DIFFERENT LURASIDONE FORMULATIONS IN PATIENTS WITH SCHIZOPHRENIA, SCHIZOAFFECTIVE, OR SCHIZOPHRENIFORM DISORDER
Brief Title: The Bioequivalence Of Two Different Lurasidone Formulations In Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: D1050263
Record Dates: First submitted 2010-03-05; First posted 2010-03-08 (Estimated); Last update posted 2011-09-08 (Estimated); Status verified 2011-09

CONDITIONS: Schizophrenia
Keywords: Bioequivalence; Male/Female Patient; Reference/Test Formulation; Schizophrenia Patients
MeSH Terms: conditions — Schizophrenia | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reference Formulation (Other): Dosed 12.5% drugload 3X40mg
  Interventions: Drug: Lurasidone HCl
- Test Formulation (Other): 25% Drugload 1X120mg
  Interventions: Drug: Lurasidone HCl

INTERVENTIONS:
Drug: Lurasidone HCl — 120mg dose. 3-way cross-over for 21 days

SUMMARY:
A Phase I, Bioequivalent Study between 2 Formulations of Lurasidone HCl

DETAILED DESCRIPTION:
12.5% Drugload 3X40mg vs. 25% Drugload 1X120mg

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of schizophrenia, schizoaffective disorder, or schizophreniform disorders as per DSM-IV or DSM-IV-TR criteria, which in the opinion of the investigator have been clinically stable for the past 6 months.
2. Body mass index (BMI) ≥ 19.5 and ≤ 37 kg/m2.
3. No clinically relevant abnormal laboratory values.
4. No clinically significant findings in the 12-lead electrocardiogram (ECG):
5. No clinically significant findings from a vital signs measurement.
6. Able to understand and provide written consent prior to initiating any study procedure after being informed of the nature of the study.
7. Females who participate in this study:

   * are unable to have children (e.g. post-menopausal, tubal ligation, hysterectomy); OR
   * are willing to remain abstinent [not engage in sexual intercourse] from Day -5 until the final follow-up visit; OR
   * are willing to use an effective method of double-barrier birth control (e.g. partner using condom and female using diaphragm, contraceptive sponge, spermicide, or intrauterine device [IUD]) from Day -5 until the final follow-up visit.
8. Males must be willing to remain sexually abstinent or use an effective method of birth control (e.g. condom) from Day -5 until the final follow-up visit.

Exclusion Criteria:

1. Significant disease(s) or clinically significant finding(s) in a physical examination determined by an Investigator to pose a health concern to the patient while on study.
2. Known history or presence of intolerance to psychiatric medications (e.g. atypical antipsychotic medications).
3. History of alcohol or drug-dependence as per DSM-IV criteria during the 6-month period immediately prior to study entry.
4. Significant orthostatic hypotension (i.e. a drop in systolic blood pressure of 30 mmHg or more and/or drop in diastolic blood pressure of 20 mmHg or more on standing).
5. Presence or history (within the last year) of a medical or surgical condition (e.g. gastrointestinal disease) that might interfere with the absorption, metabolism, or excretion of orally administered lurasidone.
6. A history of epilepsy or risk of having seizures.
7. Positive test results within 30 days prior to the start of the study for:

   1. Human immunodeficiency virus (HIV).
   2. Hepatitis B surface antigen and Hepatitis C antibody.
   3. Urine drugs of abuse test (marijuana, amphetamines, barbiturates, cocaine, opiates, benzodiazepines and methadone).
   4. Serum beta-HCG consistent with pregnancy (females only).
8. Participated in another clinical trial or received an investigational product within 30 days prior to Screening.
9. Use of any inhibitor or inducer of CYP3A4 taken within 30 days prior to check-in, including but not limited to those listed in Appendix 19.3.
10. Difficulty fasting or consuming the standard meals.
11. Females taking oral or transdermal hormonal contraceptives within 14 days preceding period 1 dosing.

    -OR- Females having used implanted or injected hormonal contraceptives within 6 months prior to period 1 dosing.
12. Donation or loss of whole blood prior to drug administration, as follows:

    1. ≤ 499 mL within 30 days prior to dosing
    2. ≥ 500 mL within 56 days prior to dosing.
13. Patient has a prolactin concentration ≥ 100 ng/mL at Screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2008-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lev Gertsik, MD, Principal Investigator — California Clinical Trials (CCT)
Locations (1):
- California Clinical Trials (CCT), Glendale, California, United States